CLINICAL TRIAL: NCT02343835
Title: IRE: Anti-Tumor Immunity Induced by IRE of Unresectable Pancreatic Cancer
Brief Title: Anti-Tumor Immunity Induced by IRE of Unresectable Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JF-20150113(4)
Record Dates: First submitted 2015-01-12; First posted 2015-01-22 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2019-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NanoKnife LEDC System (Experimental): 90 pulses of 70 microseconds each in duration will be administered per electrode pair.
  Interventions: Device: NanoKnife LEDC System
- Control (No Intervention): The patients without treatment

INTERVENTIONS:
Device: NanoKnife LEDC System — Irreversible electroporation (IRE) is a new, minimal-invasive image-guided treatment method for tumors not amenable for surgical resection or thermal ablation, due to vicinity near vital structures such as vessels and bile ducts. With IRE, multiple electrical pulses are applied to tumorous tissue. These pulses alter the existing transmembrane potential of the cell membranes, and create 'nanopores', after which the cell dies through loss of homeostasis.
  Other Names: NanoKnife
  Arms: NanoKnife LEDC System

SUMMARY:
This protocol will study the impact of Irreversible electroporation (IRE) on immune response in patients diagnosed with unresectable pancreatic cancers smaller than 5.0 cm. It will profile the immune response to IRE of unresectable pancreatic cancers. The intra-tumoral and systemic immune response to IRE will be determined and compared to pre-ablated pancreatic cancer specimens and historical control specimens.

DETAILED DESCRIPTION:
Thirty patients with histologically confirmed locally advanced pancreatic adenocarcinoma (≤5.0cm) will undergo percutaneous irreversible electroporation of the tumor using CT and ultrasound guidance. Blood will be drawn for research before IRE. Blood and tissue samples will be used.

After IRE, patients will be carefully monitored and systemic immune responses are registered. Follow-up will consist of frequent CT and MRI scanning, as well as serum CA19.9 tumor marker and quality of life questionnaires and overall survival (OS).

The investigators hypothesize that IRE in the pancreas will induce good symptom palliation without causing severe complications as well as perfect systemic immune response.

ELIGIBILITY:
Inclusion Criteria:

* Radiologic confirmation of unresectable pancreatic cancer by at least CT of chest and abdomen
* Screening must be performed no longer than 2 weeks prior to study inclusion
* Maximum tumor diameter ≤ 5 cm;
* Histological or cytological confirmation of pancreatic adenocarcinoma;
* Age ≥ 18 years;
* ASA-classification 0 - 3
* Life expectancy of at least 12 weeks;
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to definite inclusion;

  * Hemoglobin ≥ 5.6 mmol/L;
  * Absolute neutrophil count (ANC) ≥ 1,500/mm3;
  * Platelet count ≥ 100*109/l;
  * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN);
  * ALT and AST ≤ 2.5 x ULN;
  * Serum creatinine ≤ 1.5 x ULN or a calculated creatinine clearance ≥ 50 ml/min;
  * Prothrombin time or INR < 1.5 x ULN;
  * Activated partial thromboplastin time < 1.25 x ULN (therapeutic anticoagulation therapy is allowed if this treatment can be interrupted as judged by the treating physician);
* Written informed consent;

Exclusion Criteria:

* Resectable pancreatic adenocarcinoma as discussed by our multidisciplinary hepatobiliary team;
* Successful down staging after (radio)chemotherapy from previous unresectable/borderline tumor to resectable tumor;
* History of epilepsy;
* History of cardiac disease:

  * Congestive heart failure >NYHA class 2;
  * Active Coronary Artery Disease (defined as myocardial infarction within 6 months prior to screening);
  * Cardiac arrhythmias requiring anti-arrhythmic therapy or pacemaker (beta blockers for antihypertensive regimen are permitted);
* Uncontrolled hypertension. Blood pressure must be ≤160/95 mmHg at the time of screening on a stable antihypertensive regimen;
* Compromised liver function (e.g. signs of portal hypertension, INR > 1,5 without use of anticoagulants, ascites);
* Uncontrolled infections (> grade 2 NCI-CTC version 3.0);
* Pregnant. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment;
* Immunotherapy ≤ 6 weeks prior to the procedure;
* Chemotherapy ≤ 6 weeks prior to the procedure;
* Radiotherapy ≤ 6 weeks prior to the procedure;
* Concomitant use of anti-convulsive and anti-arrhythmic drugs (other than beta blockers used for antihypertensive);
* Allergy to contrast media;
* Any implanted stimulation device;
* Any implanted metal stent/device within the area of ablation that cannot be removed;
* Any condition that is unstable or that could jeopardize the safety of the subject and their compliance in the study; Of note, patients with contra-indications for MRI will not be excluded from participation: in this case radiologic follow-up will consist of CT-scanning according to protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Characterization of the intra-tumoral and systemic immune response to IRE in unresectable pancreatic cancers | 12 Months
  1. Determine number (percentage via flow cytometry), phenotype and functionality of tumor infiltrating lymphocytes in ablated pancreatic cancer
  2. Determine morphology and histology of regional lymph node after IRE
  3. Quantify T cell response (IUs of IL2 and IFN gamma, and T cell specific cells as measured by number of spots on an elispot assay) to tumor associated antigens using in vitro assays of T cell proliferation and function (cytokine release, elispot, peptide-MHC)

SECONDARY OUTCOMES:
Comparison immune response between non-ablated and ablated pancreatic cancer and pre-ablated and post ablated serum | 24 Months
  1. Compare serum cytokine and chemokine expression (in IU) between patients undergoing or not undergoing tumor ablation
  2. Characterize cytokine and chemokine expression (in IU) in ablated tissue and in pre-ablated and post-ablated serum over time
  3. Compare intra-tumoral lymphocyte populations (percentage via flow cytometry) in ablated tumor tissue with paraffin embedded specimens for tumors that are matched for age, tumor size and histology.

OTHER OUTCOMES:
Overall survival and (local and distant) progression-free survival. | 60 Months

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi l Niu, M.D.,PHD., Study Chair — FUDA Cancer Hospital
Locations (1):
- FUDA Cancer Hospital, Guangzhou, Guangdong, China